CLINICAL TRIAL: NCT04132583
Title: A Randomized, Open-label, Single Dose, Two-Treatment, Two Period Crossover Design (2x2), Comparative Bioequivalence Study of Deflox® Tablets 50 mg vs Cataflam DD ® Tablets 50 mg (Innovator) in Healthy Volunteers
Brief Title: Deflox Tablets Bioequivalence (BE) Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MS200505_0003
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: Deflox®; Cataflam® DD; Diclofenac potassium; Healthy
MeSH Terms: interventions — Terazosin; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Deflox®, Then Cataflam DD® (Experimental): Participants received single oral dose of Deflox® 50 milligrams (mg) tablet in Treatment Period 1 followed by a single oral dose of Cataflam DD® 50 mg tablet in Treatment Period 2 under fasting condition. A wash-out period of 7 days was maintained between the Treatment Periods 1 and 2.
  Interventions: Drug: Deflox®; Drug: Cataflam DD®
- First Cataflam DD®, Then Deflox® (Experimental): Participants received single oral dose of Cataflam DD® 50 mg tablet in Treatment Period 1 followed by single oral dose of Deflox® 50 mg tablet in Treatment Period 2 under fasting condition. A wash-out period of 7 days was maintained between Treatment Periods 1 and 2.
  Interventions: Drug: Deflox®; Drug: Cataflam DD®

INTERVENTIONS:
Drug: Deflox® — Participants received a single oral dose of 50 mg Deflox® tablet in either treatment period 1 or 2 under fasting conditions.
  Other Names: Diclofenac Potassium
Drug: Cataflam DD® — Participants received a single oral dose of 50 mg Cataflam DD® tablet in either treatment period 1 or 2 under fasting conditions.

SUMMARY:
The purpose of this study was to demonstrate the bioequivalence of Deflox® 50 milligrams (mg) tablets compared with Cataflam® DD tablets 50 mg administered as single dose in fasting conditions to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a body weight within 55-95 kilograms (kg) and body mass index (BMI) within the range 18.0-27.0 kilogram/meter square (kg/m2) (inclusive)
* Participant has given written informed consent before any study-related activities are carried out - Participants with ethnic origin: Mexicans (example: Caucasians, Indigenous peoples and Mestizos) - No smoking
* Participants with good physical and mental health status, determined on the basis of the medical history and a physical examination
* All values for biochemistry and hematology tests of blood and urine within the normal range or showing no clinically relevant deviation as judged by the Investigator
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with any surgical or medical condition, including findings in the medical history or in the pre-study assessments, or any other significant disease, that in the opinion of the investigator, constitutes a risk or a contraindication for the participation of the participant in the study or that could interfere with the study objectives, conduct or evaluation
* Participants with history of surgery of the gastrointestinal tract which could influence the gastrointestinal absorption and/or motility according to the Investigator's opinion
* Participants with allergy: ascertained or presumptive hypersensitivity to the active drug substance and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the trial
* A subpopulation of participants with asthma may have aspirin-sensitive asthma, which may include chronic rhinosinusitis complicated by nasal polyps; severe, potentially fatal bronchospasm; and/or intolerance to aspirin and other nonsteroidal anti-inflammatory drugs (NSAIDs). Because cross-reactivity between aspirin and other NSAIDs has been report in such aspirin-sensitive patients, Cataflam is contraindicated in patients with this form of aspirin sensitivity
* Receipt of any prescription or non-prescription medication within 2 weeks before the first study drug administration, including multivitamins and herbal products (example: St John's Wort), including acetylsalicylic acid (ASA), and hormonal contraceptives in females
* Participants with renal failure or renal dysfunction (creatinine clearance < 80 milliliter per minute [mL/min]) as assessed by using the estimated measure with the Cockcroft-Gault formula
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-21 (Actual); Primary Completion 2019-10-27 (Actual); Study Completion 2019-10-27 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Diclofenac | Pre-dose up to 24 hours Post-dose
Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of Diclofenac | Pre-dose up to 24 hours Post-dose
Maximum Observed Plasma Concentration (Cmax) of Diclofenac | Pre-dose up to 24 hours Post-dose

SECONDARY OUTCOMES:
Time to Reach Maximum Plasma Concentration (Tmax) of Diclofenac | Pre-dose up to 24 hours Post-dose
Terminal Elimination Half-Life (t1/2) of Diclofenac | Pre-dose up to 24 hours Post-dose
Apparent Volume of Distribution During Terminal Phase (Vz/f) of Diclofenac | Pre-dose up to 24 hours Post-dose
Apparent Total Body Clearance of Drug From Plasma (CL/f) of Diclofenac | Pre-dose up to 24 hours Post-dose
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs | Baseline up to 15 days (end of study)
Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters | Baseline up to 15 days (end of study)
Number of Participants With Clinically Significant Abnormalities in Vital Signs | Baseline up to 15 days (end of study)
Number of Participants With Clinically Significant Abnormalities in 12-lead Electrocardiogram (ECG) | Baseline up to 15 days (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Clinica de Enfermedades Crónicas y de Procedimientos Especiales S.C., Morelia, Mexico

IPD SHARING:
Plan to Share IPD: No
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany, will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.merckgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200505_0003
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html